CLINICAL TRIAL: NCT01329068
Title: Patient Empowerment by Group Medical Consultations in the Follow-up of Breast Cancer Survivors and Surveillance of Women With a BRCA Mutation
Brief Title: Patient Empowerment by Group Medical Consultations
Acronym: GMC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCNONCO201006
Record Dates: First submitted 2011-03-31; First posted 2011-04-05 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2011-10

CONDITIONS: Breast Cancer; BRCA Mutation
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individual consult (Active Comparator): regular individual consult
  Interventions: Behavioral: individual consult
- group medical consult (Active Comparator): regular group medical consult
  Interventions: Behavioral: group medical consult

INTERVENTIONS:
Behavioral: individual consult — regular individual consultations
  Arms: Individual consult
Behavioral: group medical consult — group medical consult
  Arms: group medical consult

SUMMARY:
Carriers of a BRCA mutation have a significantly increased risk to develop breast cancer in the course of their lives . They face a difficult choice: either a preventive removal of the breast(s) or an intensive inspection process.

After primary treatment of breast cancer, patients will be followed for 5-10 years to diagnose recurrence or a new primary tumor in an early stage; to support the patient during hormonal treatment; to educate the patient about risk factors and healthy life style; and to provide psychosocial support.

Currently, follow-up of breast cancer patients and surveillance of BRCA mutation carriers is offered in regular, one-to-one medical visits. Experience shows that in an individual visit it is often not possible to give all aspects that are important, enough attention. The group medical consultation (GMC) is a new form of medical visits where the physician or nurse practitioner performs a series of one-to-one consultations in the presence of 8 to10 other patients. A social worker accompanies this process. Patients in group consultations may gather more information because they learn from each other and there is relatively more time compared to a regular consultation. Research shows that both patients and caregivers are more satisfied with care after a group consultation compared to individual visits. After a GMC the participants from the breast cancer GMCs will be provided with a dedicated iPad for 3 months. Using this iPad, patients can contact the women they have met during the GMC as well as health care professionals by several communication channels, including virtual group meetings. This approach provides a unique combination of both social support and professional education concerning survivorship in an e-health environment.However, it is also known that group sessions may be counterproductive for some patients, for example because they are frightened by the stories of others. The goal of this study is to examine whether group visits (in combination with dedicated iPads) are beneficial to women with a BRCA mutation and for patients in follow-up after breast cancer.

ELIGIBILITY:
Inclusion Criteria:

Participants: patients in follow-up after breast cancer

* Women ≥ 18 years of age with histologically proven breast cancer.
* Primary treatment (surgery, radiotherapy, chemotherapy) completed maximally 5 years ago.

Participants: women with a BRCA mutation

* Women ≥ 25 years of age with a proven BRCA1 or BRCA2 mutation.
* Carrier of a BRCA1 or BRCA2 mutation, diagnosed maximally two years before inclusion.

Exclusion Criteria:

Participants: patients in follow-up after breast cancer

* Metastatic breast cancer
* Currently involved in a diagnostic work-up because of a suspicion of breast cancer, either primary or metastatic.
* A history of prophylactic mastectomy.
* Current psychiatric disease precluding consultations in a group.
* Insufficient command of the Dutch language to be able to follow a group discussion and/or to fill out a Dutch questionnaire

Participants: women with a BRCA mutation

* Metastatic breast cancer
* Currently involved in a diagnostic work-up because of a suspicion of breast cancer, either primary or metastatic.
* A history of prophylactic mastectomy.
* Current psychiatric disease precluding consultations in a group.
* Insufficient command of the Dutch language to be able to follow a group discussion and/or to fill out a Dutch questionnaire

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2011-04; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Psychological distress (SCL-90) and empowerment (Cancer Empowerment Questionnaire) | BRCA mutation carriers: Baseline (1 week before the (group) medical visit) and 1 week and three months after the (group) medical visit.

SECONDARY OUTCOMES:
Questionnaires for patients and health care professionals, observations and user measurements of the iPads. | BRCA mutation carriers: Baseline (1 week before the (group) medical visit) and 1 week and three months after the (group) medical visit.
  * Cancer worry (CWS)
  * Quality of life (EORTC QLQ C30 and BR23)
  * Compliance to hormonal treatment (MARS) (for breast cancer only)
  * Cost-effectiveness (TIC-P- part 1 and EuroQol-5D)
  * Information needs and giving
  * Self-breast examination (for BRCA only)
  * Decisions for prophylactic mastectomy or surveillance (for BRCA only)
  * Patient satisfaction
  IPads:
  * Frequency of using the iPad
  * Content of use
  * Frequency and ways of contacting other patients
  * Content of the online meetings

CONTACTS AND LOCATIONS:
Overall Officials: H.W.M. van Laarhoven, Md PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Visser A, Prins JB, Hoogerbrugge N, van Laarhoven HW. Group medical visits in the follow-up of women with a BRCA mutation: design of a randomized controlled trial. BMC Womens Health. 2011 Aug 24;11:39. doi: 10.1186/1472-6874-11-39. PMID 21864353